CLINICAL TRIAL: NCT06702033
Title: Phase II Trial of Surgery Followed by Risk-Directed Post-Operative Adjuvant Therapy for HPV-Related Oropharynx Squamous Cell Carcinoma: "The Minimalist Trial-2 (MINT-2)"
Brief Title: The Minimalist Trial-2
Acronym: MINT-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Joseph Sanchez Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202501127
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: HPV-Related Oropharynx Squamous Cell Carcinoma
Keywords: De-escalation; Adjuvant therapy; Oropharyngeal cancer; Human papillomavirus
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiotherapy; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: * Highest risk pathology (pT4) = remove from trial.
  * High-risk pathology = Arm 1
  * Intermediate-risk pathology will be randomized to Arm 2A, Arm 2B, or Arm 2C.
  * Low-risk pathology = remove from trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Radiation therapy + Cisplatin (Experimental): * Standard of care surgery will occur before adjuvant therapy.
  * It is recommended that radiation therapy begin within 28 to 49 days (and no later than 56 days).
  * The total dose to the postoperative tumor bed will be 4200 cGy in 21 fractions of 200 cGy each over 4 weeks.
  * Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 3780 cGy in 21 fractions of 180 cGy each.
  * Cisplatin will be given on the same day as one of the initial 5 doses of radiation therapy.
  Interventions: Radiation: Radiation therapy; Drug: Cisplatin; Procedure: Surgery
- Arm 2A: Radiation therapy (Experimental): * Standard of care surgery will occur before adjuvant therapy.
  * It is recommended that radiation therapy begin within 28 to 49 days (and no later than 56 days).
  * The total dose to the postoperative tumor bed will be 4200 cGy in 21 fractions of 200 cGy each over 4 weeks.
  * Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 3780 cGy in 21 fractions of 180 cGy each.
  Interventions: Radiation: Radiation therapy; Procedure: Surgery
- Arm 2B: Radiation therapy (Experimental): * Standard of care surgery will occur before adjuvant therapy.
  * It is recommended that radiation therapy begin within 28 to 49 days (and no later than 56 days).
  * The total dose to the postoperative tumor bed will be 3780 cGY in 21 fractions of 180 cGy each over 4 weeks.
  * Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 3360 cGy in 21 fractions of 160 cGy each.
  Interventions: Radiation: Radiation therapy; Procedure: Surgery
- Arm 2C: Radiation therapy + Cisplatin (Experimental): * Standard of care surgery will occur before adjuvant therapy.
  * It is recommended that radiation therapy begin within 28 to 49 days (and no later than 56 days).
  * The total dose to the postoperative tumor bed will be 3000 cGy in 15 fractions of 200 cGy over 3 weeks.
  * Additional regions in the ipsilateral and contralateral neck at risk for microscopic disease in the cervical lymph nodes will receive 2700 cGy in 15 fractions of 180 cGy each.
  * Cisplatin will be given on the same day as one of the initial 5 doses of radiation therapy.
  Interventions: Radiation: Radiation therapy; Drug: Cisplatin; Procedure: Surgery

INTERVENTIONS:
Radiation: Radiation therapy — IMRT or IMPT
Drug: Cisplatin — Dose of 100 mg/m^2 IVPB over 60 minutes
  Arms: Arm 1: Radiation therapy + Cisplatin; Arm 2C: Radiation therapy + Cisplatin
Procedure: Surgery — Standard of care

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is the sixth most common cancer. Oropharynx SCC (OPSCC) is a common sub-type of HNSCC. Each year, 16,000 new cases of OPSCC are diagnosed in the USA. Most cases of OPSCC (>90%) are caused by the human papillomavirus (HPV) and are often cured with current therapy.

However, patients treated with surgery followed by postoperative adjuvant chemotherapy and radiation therapy (POA(C)RT) still experience substantial morbidity. In this highly curable disease, current clinical research interest is focused on investigation of de-escalated therapy, with the goal to reduce treatment-related adverse events (AEs) while maintaining a low recurrence rate.

In this study, patients with HPV-related OPSCC will undergo resection of the primary tumor site and involved/at-risk regional neck nodes. Based on the pathology report, patients will be assigned to:

* Arm 1 (de-POACRT-42 Gy)
* Arm 2A (de-POART-42 Gy)
* Arm 2B (de-POART-37.8 Gy)
* Arm 2C (de-POACRT-30 Gy).

All patients with high-risk pathology will be assigned to Arm 1 whereas patients with intermediate-risk pathology will be randomized (1:1:1) to Arm 2A, Arm 2B, or Arm 2C. Patients with highest-risk pathology and low-risk pathology will be removed from the trial after surgery and will be advised to pursue standard of care options.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HPV-related, clinical stages I-II OPSCC (8th edition of AJCC/UICC Staging Manual) or HPV-related neck node with unknown primary. Clinical T1N0M0 and T2N0M0 disease are excluded. HPV-related may be defined by p16 IHC stain and/or HPV-High Risk RNA ISH/HPV DNA genotyping by PCR, using standard definitions of positive and negative test results.
* Planned resection of the primary tumor site by a transoral approach (TORS, TLM, or conventional surgery).
* Planned unilateral or contralateral selective neck dissection.
* ECOG PS 0-2.
* Adequate organ and marrow function defined as:

  * Creatinine clearance ≥ 50 mL/min.
  * ANC ≥ 1.0 K/cumm.
  * Platelet count ≥100 K/cumm.
* At least 18 years of age.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Clinical T1N0M0 or T2N0M0 disease.
* Prior radiation therapy for HNSCC.
* Planned free-flap reconstruction of the resected primary site.
* Cirrhosis with Child-Pugh Score B or C.
* History of prior invasive malignancy diagnosed within 2 years prior to study enrollment; exceptions are malignancies with a low risk of metastasis or death (e.g., expected 5-year OS > 90%) that were treated with curative-intent therapy.
* Receiving any other investigational agents.
* Uncontrolled serious inter-current illness or serious psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. A negative serum pregnancy test is required at screening for all female patients of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2033-07-15 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | At 2 years

SECONDARY OUTCOMES:
Percent weight loss | From start of radiation therapy to completion of radiation therapy (estimated to be 6 weeks)
  For assessing percent weight loss, weight (kg) will be collected weekly during radiation within each arm, starting at Day 1 of RT and ending on the last day of RT. The percent weight loss from the baseline is calculated at any post-baseline.
Proportion of patients undergoing PEG tube placement | Through completion of follow-up (estimated to be 5 years and 10 weeks)
Duration of need for an indwelling PEG tube | Through completion of follow-up (estimated to be 5 years and 10 weeks)
Proportion of patients taking narcotic | Through completion of follow-up (estimated to be 5 years and 10 weeks)
Number of participants with adverse events | From start of surgery through 24-month follow-up visit (estimated to be 2 years and 10 weeks)
Mean change in serum creatinine during radiation therapy | From start of radiation therapy to completion of radiation therapy (estimated to be 6 weeks)
  Serum creatinine levels are collected at Day 1 of RT and ending on the last day of RT.
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 5 years and 10 weeks)
  PFS will be calculated from the date of surgery to the date of progression, death of any cause, or last known date alive.
Overall survival (OS) | Through completion of follow-up (estimated to be 5 years and 10 weeks)
  OS will be calculated from the date of surgery to the date of death or last known date alive.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices), and the study protocol will be shared, beginning 9 months and ending 24 months following article publication, with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Types of acceptable analyses include approved proposal(s) or individual participant data for meta-analyses.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 24 months following article publication.
Access Criteria: Information regarding submitting proposals and accessing data may be submitted to jcley@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu